CLINICAL TRIAL: NCT02325388
Title: Effectiveness of a Pressure-sensing System to Reduce the Risk of Pressure Ulcer Formation by Lowering Interface Pressure in Vulnerable Patient Populations: A Parallel-two-group Randomized Controlled Trial
Brief Title: Pressure Sensing to Reduce the Risk of Pressure Ulcer Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Ward of the 21st Century (Other); Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Chester Ho, MD, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB13-0794
Record Dates: First submitted 2014-12-17; First posted 2014-12-25 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer; decubitus ulcer; bed sore; continuous pressure mapping; interface pressure imaging
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group with ForeSite PT™ system (Experimental): Inpatients assigned to the treatment group with the ForeSite PT™ system will have its LCD monitor turned on (i.e., real-time images of interface pressure will be displayed on the monitor) during their enrolment in the trial.
  Interventions: Device: ForeSite PT™ system
- Control group (No Intervention): Inpatients assigned to the control group will have the ForeSite PT™ system's LCD monitor turned off and hidden (i.e., real-time images of interface pressure will not be displayed on the monitor). As the ForeSite PT™ system will continue to record interface pressure with the display turned off, this enables patients enrolled in the control group to undergo silent monitoring.

INTERVENTIONS:
Device: ForeSite PT™ system — XSENSOR Technology Corporation's ForeSite PT™ Patient Turn System (referred to as the "ForeSite PT™ system") continuously monitors interface pressure and provides CPI that quantifies real-time interface pressure information. It also provides patient turn tracking to assist with management of the patient turn schedule by alerting healthcare providers and/or caregivers to the location of body areas that have experienced the greatest exposure, and when the next turn/repositioning is due as per pre-set alerts.
  Arms: Treatment group with ForeSite PT™ system

SUMMARY:
Pressure ulcers are prevalent conditions that result in substantial financial costs to the healthcare system as well as significant distress to affected patients and their families. This study is a parallel two-group randomized controlled trial that aims to study how the use of a pressure sensing device with continuous visual feedback of pressure imaging may potentially decrease the interface pressure of patients who are at risk of pressure ulcers in an acute hospital setting.

DETAILED DESCRIPTION:
Background: Pressure ulcers result in substantial financial costs to the healthcare system as well as significant distress to affected patients and their families. As interface pressure is a key risk factor in the development of pressure ulcers, continuous visual feedback of continuous pressure imaging (CPI) between the body and support surface could inform healthcare providers on repositioning strategies and play a key role in an overall strategy for the prevention and management of pressure ulcers. This randomized, controlled trial aims to study the effect of CPI on the reduction of interface pressure, and the incidence of pressure ulcers in vulnerable hospital patients.

Methods: A parallel two-group randomized controlled clinical trial will be conducted. A total of 678 eligible consenting inpatients at high risk of pressure ulcer development in a tertiary acute care institution will be randomly allocated to either have the ForeSite PT™ system with the liquid-crystal display ("LCD") monitor turned on to provide visual feedback through CPI to healthcare providers while also collecting continuous interface pressure data (intervention group), or have the ForeSite PT™ system with the LCD monitor turned off, therefore not providing visual feedback or CPI to healthcare providers, while collecting continuous interface pressure data in the background (control group), in a ratio of 1:1. Data will be collected on both groups for three days (72 hours). The primary outcome will be the differences in the two groups' interface pressure analysis. The interface pressure readings will be collected through hourly sampling of continuous interface pressure recordings taken throughout this study period. Clinical outcomes will be the differences in the two groups' pressure-related skin and soft tissue change in areas at risk of pressure ulcer. It will be obtained at baseline (within 24 hours of admission) and on the third day of the trial. Perceptions of intervention patients and healthcare providers will be obtained on the third day.

Discussion: This will be the first randomized controlled trial to investigate the effect of CPI on interface pressure of vulnerable hospital patients, and the association between interface pressure and development of pressure-related skin and soft tissue changes. The results could provide important information to guide clinical practice in the prevention and management of pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adult, man or woman, with a minimum age limit of 18 years old.
* Expected to have a length of stay on the unit of at least three days.
* Require assistance with bed mobility or completely dependent for bed mobility as determined by the "Bed" components in the de Morton Mobility Index (DEMMI). Eligible patients would be:

  1. Unable (score of "0") to bridge, roll onto their side, and sit from lying supine.
  2. Unable (score of "0") to bridge and roll onto their side, and requires minimal assistance and/or supervision with sitting from lying supine.
  3. Able (score of "1") to bridge, unable to roll onto their side (score of "0"), and requires minimal assistance and/or supervision with sitting from lying supine.
* Capacity to provide consent, or have a surrogate decision-maker provide consent on their behalf.
* Not near the end of life within three days of enrolment in the study.

Exclusion Criteria:

* Have a planned admission to another unit (including those identified as a setting for data collection in the study) within three days of enrolment in the study.
* Sleep in a chair at night.
* Whose clinical care would be negatively impacted if turned or repositioned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2014-12; Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Interface pressure analysis - peak pressure | 72 hours
  Peak pressure of any given pressure reading sample
Interface pressure analysis - sensel pressure reading | 72 hours
  Absolute number of sensels with pressure readings greater than 40 mmHg
Interface pressure analysis - average pressure | 72 hours
  Average interface pressure (excluding sensels with 0mmHg reading)
Interface pressure analysis - % with pressure over 40mmHg | 72 hours
  Proportion of participants that have pressure readings greater than 40 mmHg

SECONDARY OUTCOMES:
Pressure related skin and soft tissue changes | 72 hours
  Any change in the skin appearance, pressure ulcer formation, skin/wound infection
Perceptions of healthcare providers | 72 hours
  Survey of healthcare providers on prior experience with pressure mapping technology, functionality, ease of use, and interpretation of pressure data on the LCD monitor.
Perceptions of patients | 72 hours
  Survey of patients on prior and current experience with CPI (including sensor mattress cover and monitor display of their pressure distribution) on their care and comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Chester H Ho, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ho C, Ocampo W, Southern DA, Sola D, Baylis B, Conly JM, Hogan DB, Kaufman J, Stelfox HT, Ghali WA. Effect of a Continuous Bedside Pressure Mapping System for Reducing Interface Pressures: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2316480. doi: 10.1001/jamanetworkopen.2023.16480. PMID 37266939
- [Derived] Wong H, Kaufman J, Baylis B, Conly JM, Hogan DB, Stelfox HT, Southern DA, Ghali WA, Ho CH. Efficacy of a pressure-sensing mattress cover system for reducing interface pressure: study protocol for a randomized controlled trial. Trials. 2015 Sep 29;16:434. doi: 10.1186/s13063-015-0949-x. PMID 26420303